CLINICAL TRIAL: NCT01436500
Title: A Multi-Center, Double-Blind, Randomized, Controlled Study to Determine the Safety and Pharmacokinetics of Ifetroban Injection in Hepatorenal Syndrome
Brief Title: Safety and Pharmacokinetics of Ifetroban in Hepatorenal Syndrome Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPI-IFE-001
Record Dates: First submitted 2011-08-31; First posted 2011-09-19 (Estimated); Results first posted 2017-02-14 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Hepatorenal Syndrome
Keywords: Hepatorenal Syndrome; HRS; ifetroban
MeSH Terms: conditions — Hepatorenal Syndrome | interventions — ifetroban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- 5 mg ifetroban, Type 1 (Experimental): 60-minute intravenous infusion of 5 mg ifetroban given once daily for 3 days to subjects with Type 1 HRS.
  Interventions: Drug: Ifetroban Injection
- Placebo, Type 1 (Placebo Comparator): 60-minute intravenous infusion of 5% dextrose in sterile water given once daily for 3 days to subjects with Type 1 HRS.
  Interventions: Drug: Placebo
- 5 mg ifetroban, Type 2 (Experimental): 60-minute intravenous infusion of 5 mg ifetroban given once daily for 3 days to subjects with Type 1 HRS.
  Interventions: Drug: Ifetroban Injection
- 15 mg ifetroban, Type 1 (Experimental): 60-minute intravenous infusion of 15 mg ifetroban given once daily for 3 days to subjects with Type 1 HRS.
  Interventions: Drug: Ifetroban Injection
- 15 mg ifetroban, Type 2 (Experimental): 60-minute intravenous infusion of 15 mg ifetroban given once daily for 3 days to subjects with Type 2 HRS.
  Interventions: Drug: Ifetroban Injection
- 50 mg ifetroban, Type 1 (Experimental): 60-minute intravenous infusion of 50 mg ifetroban given once daily for 3 days to subjects with Type 1 HRS.
  Interventions: Drug: Ifetroban Injection
- 50 mg ifetroban, Type 2 (Experimental): 60-minute intravenous infusion of 50 mg ifetroban given once daily for 3 days to subjects with Type 2 HRS.
  Interventions: Drug: Ifetroban Injection
- 150 mg ifetroban, Type 2 (Experimental): 60-minute intravenous infusion of 150 mg ifetroban given once daily for 3 days to subjects with Type 2 HRS.
  Interventions: Drug: Ifetroban Injection
- Placebo, Type 2 (Placebo Comparator): 60-minute intravenous infusion of 5% dextrose in sterile water given once daily for 3 days to subjects with Type 2 HRS.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ifetroban Injection — Ifetroban sodium injectable, diluted in sterile water with 5% dextrose
  Arms: 15 mg ifetroban, Type 1; 15 mg ifetroban, Type 2; 150 mg ifetroban, Type 2; 5 mg ifetroban, Type 1; 5 mg ifetroban, Type 2; 50 mg ifetroban, Type 1; 50 mg ifetroban, Type 2
Drug: Placebo — Sterile water with 5% Dextrose
  Other Names: D5W
  Arms: Placebo, Type 1; Placebo, Type 2

SUMMARY:
A study of ifetroban in the treatment of hepatorenal syndrome (HRS) in hospitalized adult patients to assess the safety and pharmacokinetics of 3 days of intravenous ifetroban.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic liver disease, defined as cirrhosis with ascites based on clinical findings (biopsy not necessary).
2. Subjects with either Type 1 or Type 2 HRS defined in a and b below:

   a. Type 1: i. At least a doubling of the serum creatinine to a minimum of 220 µmol/L (2.5 mg/dL) at enrollment, occurring over a period of less than 14 days, OR ii. A 50% or greater reduction in the estimated glomerular filtration rate (GFR - calculated by the method of Cockcroft-Gault) to below 20 mL/min at enrollment occurring over a period of less than 14 days.

   iii. A projected doubling of serum creatinine to a minimum of 2.5 mg/dL, expected to occur in less than 14 days based on the rate of change observed.

   b. Type 2: defined as at least a 33% reduction in creatinine clearance occurring over a period of greater than 2 weeks, with a serum creatinine (SCr) > 133µmol/L (1.5 mg/dL).
3. Oliguria occurring within 48 hours prior to the first administration CTM. Oliguria is defined as an average urine output of < 35 mL/hr (measured for a minimum of 4 hours) under either of the following circumstances:

   a. When measured central venous pressure (CVP) > 12 mmHg, OR b. following a fluid challenge consisting of either: i. at minimum 20 mL/kg isotonic fluid (e.g. any combination of 5% albumin, normal saline, blood or blood products) given over no more than 6 hours ii. at minimum 1 g/kg of hypertonic fluid (e.g. 25% albumin) given over no more than 24 hours iii. an equivalent combination of 3.b.i and 3.b.ii

Exclusion Criteria:

1. History of allergy or hypersensitivity to ifetroban
2. Pregnant or nursing
3. Less than 18 years of age
4. Serum creatinine at the time of enrollment greater than or equal to 5.0 mg/dL
5. Platelet count at screening less than 30 x 10^3 platelets/µL
6. Anticipated of planned need for dialysis within 5 days of first CTM dose.
7. Active gastrointestinal hemorrhage (where active is defined as evidence of bleeding within 48 hours of the first dose of CTM)
8. Evidence of current (within past 30 days) obstructive (post-renal) or intrinsic renal disease [including but not limited to: acute tubular necrosis (ATN), glomerular diseases/glomerulonephritis, acute interstitial nephritis (AIN), known urinary obstruction, proteinuria > 500 mg/day, microhematuria (> 50 RBCs/high power field), abnormal renal ultrasound, fractional excretion of sodium (FeNa) > 2.0%, any urinary casts other than hyaline.
9. Current or recent (within the preceding 5 days) treatment with nephrotoxic drugs including but not limited to: NSAIDs (prior 48 hours), angiotensin converting enzyme (ACE) inhibitors, angiotensin receptor blockers (ARB), calcineurin inhibitors (cyclosporine, tacrolimus), aminoglycosides, amphotericin B, antiretrovirals and antivirals (adefovir, cidofovir, tenofovir, acyclovir, indinavir), cisplatin, methotrexate, cyclosporine, amphotericin B contrast agents, foscarnet, zoledronate, etc.
10. Presence of shock defined as hypotension, with a mean arterial pressure less than 50 mmHG.
11. New York Heart Association class 3 or 4 heart failure.
12. Presence of hepatocellular carcinoma not transplantable by Milan criteria
13. Cardiopulmonary arrest without full recovery of mental status
14. Moribund and death expected within five days
15. Bacterial or fungal infections which have been unresponsive to at least 24 hours of appropriate antimicrobial therapy
16. Burns > 30% body surface area
17. Exposed to investigational drugs within 30 days before 1st CTM administration.
18. Inability to understand the requirements of the study. (Subjects must be willing to provide written informed consent or consent of legally recognized representative, as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB], and agree to abide by the study restrictions. If the subject is incapacitated, informed consent will be sought from a legally recognized representative).
19. Refusal to provide written authorization for use and disclosure of protected health information.
20. Be otherwise unsuitable for the study, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brendan McGuire, MD, Principal Investigator — University of Alabama at Birmingham
Locations (12):
- United States (11):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - UCSD, Hillcrest Medical Center Hospital, La Jolla, California
  - UCSF (University of California-San Francisco), San Francisco, California
  - Emory University Hospital, Atlanta, Georgia
  - Indiana University (Division of Gastroenterology/Hepatology), Indianapolis, Indiana
  - University of Michigan Hospital, Ann Arbor, Michigan
  - NYU Langone Medical Center, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Baylor All Saints Medical Center, Fort Worth, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
- MIDAS Multispeciality Hospital PVT LTD, Nagpur, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 mg Ifetroban: 5 mg Ifetroban Injection administered IV over 60 minutes once daily x 3 days
- 15 mg Ifetroban: 15 mg Ifetroban Injection administered IV over 60 minutes once daily x 3 days
- 50 mg Ifetroban: 50 mg Ifetroban Injection administered IV over 60 minutes once daily x 3 days
- 150 mg Ifetroban: 150 mg Ifetroban Injection administered IV over 60 minutes once daily x 3 days
- Placebo: 5% Dextrose in Water administered IV over 60 minutes once daily x 3 days
Period: Overall Study
Arm/Group | 5 mg Ifetroban | 15 mg Ifetroban | 50 mg Ifetroban | 150 mg Ifetroban | Placebo
Started | 12 | 12 | 12 | 6 | 13
Completed | 9 | 9 | 7 | 5 | 9
Not Completed | 3 | 3 | 5 | 1 | 4
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0
Not completed — liver transplant | 1 | 0 | 0 | 0 | 0
Not completed — initiation of dialysis | 0 | 0 | 0 | 0 | 1
Not completed — discontinued study drug | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ifetroban Injection: 5, 15, 50, or 150 mg Ifetroban Injection administered IV over 60 minutes once daily x 3 days
- Total: Total of all reporting groups
Arm/Group | Ifetroban Injection | Placebo | Total
Number analyzed (Participants) | 42 | 13 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9.7) | 56 (6.4) | 57 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 5 | 22
  Male | 25 | 8 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 34 | 7 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 37 | 12 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Half-life (T-1/2) of Ifetroban and Ifetroban Acylglucuronide
Description: Plasma concentrations of ifetroban and its major active metabolite were measured at Baseline and Study Hours 1, 2, 4, 8, 12, 24, 48, 49, 50, 52, 56, 60, and 72 to determine the Pharmacokinetic parameters.
Time Frame: 3 days
Population: Patients from which a full series of plasma samples were obtained from baseline through Hour 72 were included in the calculations of the PK parameters. Where the number of participants analyzed in an arm is lower than the number exposed for that arm, the patients with missing data did not contribute to the calculation of the PK parameters.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 5 mg Ifetroban, Type 1 | 5 mg Ifetroban, Type 2 | 15 mg Ifetroban, Type 1 | 15 mg Ifetroban, Type 2 | 50 mg Ifetroban, Type 1 | 50 mg Ifetroban, Type 2 | 150 mg Ifetroban, Type 2
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 3 | 5 | 3
hours
  half-life ifetroban: number analyzed (Participants) | 2 | 5 | 5 | 5 | 3 | 5 | 3
  half-life ifetroban | 36.0 (NA) — No SD available with a sample of 2. | 11.9 (18.4) | 15.7 (16.7) | 10.5 (8.6) | 18.1 (14.8) | 13.5 (8.2) | 17.4 (11.7)
  half-life ifetroban acylglucuronide | 17.1 (17.5) | 14.7 (19.9) | 22.1 (9.5) | 18.6 (10.9) | 26.4 (22.0) | 15.2 (9.5) | 12.6 (12.4)

2. Primary Outcome: Pharmacokinetic Parameters (Exposure) of Ifetroban and Ifetroban Acylglucuronide After Three Days of Treatment
Description: Plasma concentrations of ifetroban and its primary active metabolite were measured at Baseline and Study Hours 1, 2, 4, 8, 12, 24, 48, 49, 50, 52, 56, 60, and 72 to determine the Pharmacokinetic parameters.
Time Frame: 3 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | 5 mg Ifetroban, Type 1 | 5 mg Ifetroban, Type 2 | 15 mg Ifetroban, Type 1 | 15 mg Ifetroban, Type 2 | 50 mg Ifetroban, Type 1 | 50 mg Ifetroban, Type 2 | 150 mg Ifetroban, Type 2
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 3 | 5 | 3
ng*hr/mL
  Ifetroban area under the curve (AUC) to 24 hours | 964 (683) | 779 (326) | 2025 (639) | 2463 (1497) | 5151 (3579) | 6634 (2166) | 18612 (8408)
  Ifetroban AUC to infinity: number analyzed (Participants) | 2 | 5 | 5 | 5 | 3 | 5 | 3
  Ifetroban AUC to infinity | 2476 (NA) — Only 2 subjects were deemed evaluable for this analysis by the pharmacokineticist and SD cannot be calculated with a sample size of 2. | 906 (481) | 2959 (1941) | 3259 (2866) | 6505 (4032) | 8204 (3461) | 24657 (13425)
  Ifetroban acylglucuronide AUC to 24 hours to | 4371 (2050) | 4145 (781) | 12192 (2102) | 12038 (2734) | 46455 (2906) | 42051 (18567) | 109915 (32895)
  Ifetroban acylglucuronide AUC to infinity | 8440 (8730) | 6128 (3721) | 21962 (7404) | 29857 (27688) | 86457 (44928) | 61673 (25672) | 144951 (61311)

3. Primary Outcome: Pharmacokinetic Parameters (Concentration) of Ifetroban and Ifetroban Acylglucuronide After Three Days of Treatment
Description: Plasma concentrations of ifetroban and it's major active metabolite were measured at Baseline and Study Hours 1, 2, 4, 8, 12, 24, 48, 49, 50, 52, 56, 60, and 72 to determine the Pharmacokinetic parameters.
Time Frame: 3 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 5 mg Ifetroban, Type 1 | 5 mg Ifetroban, Type 2 | 15 mg Ifetroban, Type 1 | 15 mg Ifetroban, Type 2 | 50 mg Ifetroban, Type 1 | 50 mg Ifetroban, Type 2 | 150 mg Ifetroban, Type 2
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 3 | 5 | 3
ng/mL
  Minimum Concentration Ifetroban | 1.8 (4.1) | 3.4 (4.0) | 14.1 (22.6) | 23.5 (33.7) | 43.3 (36.2) | 51.1 (44.5) | 150.0 (115.5)
  Maximum Concentration Ifetroban | 483 (445) | 251 (107) | 581 (114) | 785 (225) | 1666 (1478) | 2599 (838) | 6790 (2777)
  Minimum Concentration Ifetroban Acylglucuronide | 78.4 (56.7) | 41.4 (33.1) | 241.9 (89.0) | 200.2 (114.3) | 778.0 (583.2) | 632.9 (302.9) | 1755.0 (792.4)
  Maximum Concentration Ifetroban Acylglucuronide | 384 (103) | 448 (101) | 912 (194) | 1214 (255) | 4737 (543) | 4666 (1748) | 10447 (2113)

4. Secondary Outcome: Safety: Day 28 Mortality
Time Frame: 28 days
Measure: Number; unit: percentage of participants
Arm/Group | Ifetroban Injection | Placebo
Number analyzed (Participants) | 42 | 13
percentage of participants | 17 | 15

5. Secondary Outcome: Percentage of Patients Achieving a Treatment-period Serum Creatinine Reduction Below 1.5 mg/dL
Time Frame: Day 0 through Day 5
Measure: Number; unit: percentage of participants
Arm/Group | Ifetroban Injection | Placebo
Number analyzed (Participants) | 42 | 13
percentage of participants | 21 | 15

6. Secondary Outcome: The Percentage of Patients Achieving a Reduction of Creatinine Clearance to Below Baseline on Two Consecutive Daily Measurements
Time Frame: Day 0 to Day 5
Measure: Number; unit: percentage of participants
Arm/Group | Ifetroban Injection | Placebo
Number analyzed (Participants) | 42 | 13
percentage of participants | 62 | 77

7. Secondary Outcome: Change in 24-hour Urine Volume
Description: The volume of urine collected in a 24-hour post-treatment period minus the volume collected in a 24-hour pre-treatment period.
Time Frame: Baseline to Hour 96
Population: Data were missing for the post-treatment urine volume measurements in 9 of 42 ifetroban patients and 3 of 13 placebo patients so they were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ifetroban Injection | Placebo
Number analyzed (Participants) | 33 | 10
mL | 267.3 (613.3) | -118.5 (452.2)

ADVERSE EVENTS:
Time Frame: Day 0 through Day 28
Description: A secondary objective of the study was to evaluate the tolerability and safety of ifetroban in HRS patients. All ifetroban patients are grouped together for comparison to all placebo patients for the purpose of maximizing the significance of the evaluation.
Groups:
- Ifetroban: 5, 15, 50 or 150 mg Ifetroban Injection administered IV over 60 minutes once daily x 3 days
Arm/Group | Ifetroban | Placebo
All-Cause Mortality (participants affected / at risk) | 7/42 | 2/13
Serious Adverse Events (participants affected / at risk) | 21/42 | 8/13
Other Adverse Events (participants affected / at risk) | 25/42 | 5/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ifetroban (N=42) | Placebo (N=13)
hyperglycaemia (Endocrine disorders) | 0 | 1
worsening ascites (Gastrointestinal disorders) | 0 | 1
haematemesis (Gastrointestinal disorders) | 1 | 0
haematochezia (Gastrointestinal disorders) | 1 | 0
peritoneal haemorrhage (Gastrointestinal disorders) | 2 | 0
catheter site haemorrhage (General disorders) | 1 | 0
device failure (General disorders) | 1 | 0
chronic hepatic failure (Hepatobiliary disorders) | 3 | 0
hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
hepatorenal syndrome (Hepatobiliary disorders) | 1 | 1
liver disorder (Hepatobiliary disorders) | 1 | 0
bacteraemia (Infections and infestations) | 1 | 0
peritonitis bacterial (Infections and infestations) | 1 | 0
pneumonia (Infections and infestations) | 0 | 1
complications of transplanted liver (Injury, poisoning and procedural complications) | 1 | 0
post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Blood Creatinine Increased (Investigations) | 0 | 1
mental status changes (Psychiatric disorders) | 0 | 1
renal failure (Renal and urinary disorders) | 1 | 0
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
deep vein thrombosis (Vascular disorders) | 1 | 0
shock haemorrhagic (Vascular disorders) | 1 | 0
subarachnoid haemorrhage (Vascular disorders) | 0 | 1
upper gastrointestinal haemorrhage (Vascular disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ifetroban (N=42) | Placebo (N=13)
abdominal pain (Gastrointestinal disorders) | 4 | 0
Dyspnoea (Cardiac disorders) | 5 | 0
atrial fibrillation (Cardiac disorders) | 3 | 0
chronic hepatic failure (Hepatobiliary disorders) | 3 | 0
nausea (Gastrointestinal disorders) | 3 | 0
anaemia (Blood and lymphatic system disorders) | 3 | 0
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 1
INR increased (Investigations) | 0 | 1
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
worsening renal function (Renal and urinary disorders) | 1 | 1
hypotension (Vascular disorders) | 3 | 1
worsening coagulopathy (Blood and lymphatic system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can publish data generated at their study site after multi=center study data have already been published, or after 18 months have elapsed following database lock. The sponsor may review manuscripts before submission and delay publication by an additional 60 days, if necessary.